CLINICAL TRIAL: NCT05875454
Title: Assessment of Podocyts Integrity in Glomerular Diseases.
Brief Title: Podocyts Integrity in Glomerular Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Salah Rashed, principle investigator, Assiut University
Other Study IDs: podocytes in glomeruli
Record Dates: First submitted 2023-04-30; First posted 2023-05-25 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Glomerular Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Renal biopsies fixed in formalin from patients with suspected medical renal disease will be processed and examined for histopathological diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Histopathological examination of tru-cut needle biopsy — Renal biopsies fixed in formalin from patients with suspected medical renal disease will be processed and examined for histopathological diagnosis.

SUMMARY:
* To assess the density and ultrastructural morphology of podocytes in different glomerular diseases.
* Correlate the podocyte density and ultrastuctural morphology with laboratory data, the histopathological diagnosis and the active and chronic histopathological lesions in the biopsy.

DETAILED DESCRIPTION:
Glomerular diseases are common causes of end-stage renal failure. Increasing evidence suggests that these glomerulopathies are frequently caused by primary lesions in the renal podocytes. Podocytes are highly specialized glomerular epithelial cells that form the glomerular filtration barrier together with the fenestrated endothelium and the glomerular basement membrane. The podocyte cell body bulges into the urinary space and gives long processes that branch into foot processes, enwrapping the glomerular capillaries. Adjacent podocytes interdigitate with each other at their foot processes which are bridged with a specialized intercellular junction called a slit diaphragm, which is evenly spaced areas covered by slit diaphragm proteins that facilitate podocyte-to-podocyte contact.

Podocytes live under various stresses and pathological stimuli. They adapt to maintain homeostasis, but excessive stress leads to maladaptation and injury. Podocyte injury causes proteinuria, ranging from albuminuria to massive nephrotic syndrome. The integrity of podocytes and their interaction with the glomerular basement membrane is crucial for maintenance of the intact glomerular filtration barrier. Alteration of the intercellular junctions and cytoskeletal structure of podocytes or their detachment from the membrane results in the development of albuminuria. Podocyte density is one of the best predictors of the progression in glomerular diseases. The number of podocytes seems to be very critical for kidney health as the loss of podocytes results in glomerular damage. Thus, the extent of podocyte damage and loss seems to define the progression rate in many kidney disease.

As podocytes have limited ability to repair and/or regenerate, the extent of podocyte injury is a major prognostic determinant in glomerular diseases. Therapies aimed at preventing or limiting podocyte injury and/or at promoting podocyte repair or regeneration therefore have major potential benefits. Podocytes display a remarkable ability to recover from complete effacement and to re-form interdigitating foot processes and intact slit diaphragms after pharmacological intervention.

Podocytes are the main sites of expression of the wilm's tumor suppressor gene, WT1, in the adult. WT1 is a complex gene, which plays an essential role in renal development by controlling the process of mesenchymal to epithelial transition that form the nephron. Adult podocyte maintains both epithelial and mesenchymal features and continue to express high levels of WT1. Several lines of evidence suggest that WT1 may indeed play an important role in the maintenance of normal podocyte function. Mutations in Wilms' tumor 1 cause a wide spectrum of renal manifestations, eventually leading to end-stage kidney failure. WT1 mutations have been found to cause up to 12 % of steroid resistant nephrotic syndrome in children and young adults, particularly in phenotypic females.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing renal biopsy and diagnosed as glomerular disease.

Exclusion Criteria:

* Patients diagnosed as tubule-interstitial diseases.

Ages: 10 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected to have medical renal disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
assessment of podocytes integrity in different glomerular disaeses. | 14 months
  Assessment of podocytes density which will be detected by immunohistochemical expression of WT-1 in different glomerular diseases.
  Correletion between the podocytes density with laboratory data of the cases and the histopathological diagnosis.

REFERENCES:
- [Background] Guo JK, Menke AL, Gubler MC, Clarke AR, Harrison D, Hammes A, Hastie ND, Schedl A. WT1 is a key regulator of podocyte function: reduced expression levels cause crescentic glomerulonephritis and mesangial sclerosis. Hum Mol Genet. 2002 Mar 15;11(6):651-9. doi: 10.1093/hmg/11.6.651. PMID 11912180
- [Background] Barutta F, Bellini S, Gruden G. Mechanisms of podocyte injury and implications for diabetic nephropathy. Clin Sci (Lond). 2022 Apr 14;136(7):493-520. doi: 10.1042/CS20210625. PMID 35415751
- [Background] Sever S. Role of actin cytoskeleton in podocytes. Pediatr Nephrol. 2021 Sep;36(9):2607-2614. doi: 10.1007/s00467-020-04812-z. Epub 2020 Nov 13. PMID 33188449
- [Background] Kravets I, Mallipattu SK. The Role of Podocytes and Podocyte-Associated Biomarkers in Diagnosis and Treatment of Diabetic Kidney Disease. J Endocr Soc. 2020 Mar 5;4(4):bvaa029. doi: 10.1210/jendso/bvaa029. eCollection 2020 Apr 1. PMID 32232184
- [Background] Nagata M. Podocyte injury and its consequences. Kidney Int. 2016 Jun;89(6):1221-30. doi: 10.1016/j.kint.2016.01.012. Epub 2016 Mar 19. PMID 27165817
- [Background] Dong L, Pietsch S, Englert C. Towards an understanding of kidney diseases associated with WT1 mutations. Kidney Int. 2015 Oct;88(4):684-90. doi: 10.1038/ki.2015.198. Epub 2015 Jul 8. PMID 26154924
- [Background] Lal MA, Patrakka J. Understanding Podocyte Biology to Develop Novel Kidney Therapeutics. Front Endocrinol (Lausanne). 2018 Jul 23;9:409. doi: 10.3389/fendo.2018.00409. eCollection 2018. PMID 30083135
- [Background] Mathieson PW. The podocyte as a target for therapies--new and old. Nat Rev Nephrol. 2011 Nov 1;8(1):52-6. doi: 10.1038/nrneph.2011.171. PMID 22045242
- [Background] Muller-Deile J, Schiffer M. Podocyte directed therapy of nephrotic syndrome-can we bring the inside out? Pediatr Nephrol. 2016 Mar;31(3):393-405. doi: 10.1007/s00467-015-3116-4. Epub 2015 May 5. PMID 25939817
- [Background] Testagrossa L, Azevedo Neto R, Resende A, Woronik V, Malheiros D. Immunohistochemical expression of podocyte markers in the variants of focal segmental glomerulosclerosis. Nephrol Dial Transplant. 2013 Jan;28(1):91-8. doi: 10.1093/ndt/gfs325. Epub 2012 Aug 1. PMID 22859792